CLINICAL TRIAL: NCT00695435
Title: Evaluation of Tobramycin Tear Concentrations of TOBRADEX® Ophthalmic Suspension, Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension Versus TOBREX® Ophthalmic Solution in Normal Volunteers
Brief Title: Tobramycin Tear Concentrations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Michael Brubaker, Alcon
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-08-33
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Results first posted 2010-02-05 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Dry Eye
Keywords: normal volunteers; anti-infective; tobramycin
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Tobramycin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension (Experimental): Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension
  Interventions: Drug: Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension
- TOBREX® Ophthalmic Solution (Active Comparator): TOBREX® Ophthalmic Solution
  Interventions: Drug: TOBREX Ophthalmic Solution
- TOBRADEX® Ophthalmic Suspension (Active Comparator): TOBRADEX® Ophthalmic Suspension
  Interventions: Drug: TOBRADEX Ophthalmic Suspension

INTERVENTIONS:
Drug: TOBRADEX Ophthalmic Suspension — TOBRADEX Ophthalmic Suspension 1 drop each eye at baseline
  Arms: TOBRADEX® Ophthalmic Suspension
Drug: Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension — Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension 1 drop each eye at baseline
  Arms: Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension
Drug: TOBREX Ophthalmic Solution — TOBREX Ophthalmic Solution 1 drop each eye at baseline
  Arms: TOBREX® Ophthalmic Solution

SUMMARY:
To evaluate the Tobramycin tear concentration values of TOBRADEX® Ophthalmic Suspension, Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension versus TOBREX® Ophthalmic Solution in normal volunteers.

ELIGIBILITY:
Inclusion:

* Visual Acuity (VA) of 0.6 logMAR or better
* Tear meniscus height of ≥ 0.3mm at Visit 1.
* No concomitant topical ocular medications, including artificial tears, during the study period

Exclusion

* ocular hypertension, iritis or uveitis, glaucoma
* ocular surgery, intraocular surgery or ocular laser procedures in either eye within the past six months
* epithelial herpes simplex (dendritic keratitis); Vaccinia, active or recent varicella viral disease of the cornea and/or conjunctiva; ocular Rosacea; Mycobacterial infection of the eye; and / or fungal disease of the eye
* lacrimal duct obstruction, dry eye, ocular allergies.
* contact lens within 7 days of Visit 1.
* ocular medications within 14 days of Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, single center (Alcon Eye Clinic),
Pre-assignment Details: Treatment randomization schedules were generated and maintained by the Alcon SAS Programming group. Only when the data were verified and validated and the database locked were the appropriate personnel unmasked.
Groups:
- TOBRADEX, Then Tob 0.3%/Dex 0.05%, Then TOBREX: Patients received TOBRADEX first, then Tob 0.3%/Dex 0.05%, then TOBREX
- Tob 0.3%/Dex 0.05%, Then TOBREX, Then TOBRADEX: Patients received Tob 0.3%/Dex 0.05% first, then TOBREX, then TOBRADEX
- TOBREX, Then TOBRADEX, Then Tob 0.3%/Dex 0.05%: Patients received TOBREX first, then TOBRADEX, then Tob 0.3%/Dex 0.05%
Period: Overall Study
Arm/Group | TOBRADEX, Then Tob 0.3%/Dex 0.05%, Then TOBREX | Tob 0.3%/Dex 0.05%, Then TOBREX, Then TOBRADEX | TOBREX, Then TOBRADEX, Then Tob 0.3%/Dex 0.05%
Started | 7 | 7 | 7
Completed | 7 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Overall Study
Arm/Group | Overall Study
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Tobramycin Tear Concentration Cmax (Maximum Concentration)
Description: Tear samples were collected to measure tobramycin concentrations at 2, 4, 6, 12, and 18 minutes post-drop instillation in each subject's right eye for each treatment period.
Time Frame: 2, 4, 6, 12, and 18 minutes
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension | TOBREX® Ophthalmic Solution | TOBRADEX® Ophthalmic Suspension
Number analyzed (Participants) | 21 | 21 | 21
µg/mL | 853 (618) | 527 (428) | 542 (425)

2. Secondary Outcome: Tobramycin Tear Concentration Area Under the Curve (AUC)
Description: Trapezoidal AUC was calculated from 2 to 18 minutes.
Time Frame: 2 to 18 minutes post administration
Measure: Mean (Standard Deviation); unit: min*ug/mL
Arm/Group | Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension | TOBREX® Ophthalmic Solution | TOBRADEX® Ophthalmic Suspension
Number analyzed (Participants) | 21 | 21 | 21
min*ug/mL | 6124 (4776) | 2119 (1820) | 2484 (2182)

ADVERSE EVENTS:
Groups:
- TOBREX®: TOBREX® Ophthalmic Solution
- TOBRADEX®: TOBRADEX® Ophthalmic Suspension
Arm/Group | Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension | TOBREX® | TOBRADEX®
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tobramycin 0.3% / Dexamethasone 0.05% Ophthalmic Suspension (N=21) | TOBREX® (N=21) | TOBRADEX® (N=21)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes